CLINICAL TRIAL: NCT01464307
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Multi-center Study With an Open-label Extension Period to Investigate the Efficacy and Safety of NT 201 in the Treatment of Post-stroke Spasticity of the Lower Limb
Brief Title: Efficacy and Safety Study of Botulinum Toxin Type A Against Placebo to Treat Spasticity in the Leg After a Stroke
Acronym: PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ 60201/SP/3002; 2010-024579-23 (EudraCT Number)
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Post-stroke Spasticity of the Lower Limb
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IncobotulinumtoxinA (Xeomin) 400 Units (Experimental): IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  Interventions: Drug: IncobotulinumtoxinA (400 Units)
- Placebo Comparator Arm (Placebo Comparator): Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: IncobotulinumtoxinA (400 Units) — Main period: One injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400 units, total volume 8.0 mL; Mode of administration: intramuscular injection.
  Arms: IncobotulinumtoxinA (Xeomin) 400 Units
Drug: Placebo Comparator — Main period: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding total placebo volume 8.0 mL; Mode of administration: intramuscular injection
  Arms: Placebo Comparator Arm

SUMMARY:
The purpose of this study is to determine whether injections of Botulinum toxin type A into muscles of the leg are effective in treating patients with increased muscle tension/uncontrollable muscle stiffness (spasticity) after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-80 yrs
* Lower limb spasticity
* Time since stroke greater than 3 months
* Need for 400 U Botulinum toxin type A

Exclusion Criteria:

* Body weight below 50kg
* Fixed contractures of the lower limb
* Generalized disorders of muscle activity like Myasthenia gravis that preclude use of Botulinum toxin type A
* Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (53):
- United States (12):
  - Merz Investigational Site #001184, Downey, California
  - Merz Investigational Site #001208, Long Beach, California
  - Merz Investigational Site #001244, Fairfield, Connecticut
  - Investigational site #001188, Doral, Florida
  - Merz Investigational Site # 001110, Overland Park, Kansas
  - Merz Investigational Site #001209, Columbia, Missouri
  - Merz Investigational Site #001210, St Louis, Missouri
  - Merz Investigational Site #001198, Stratford, New Jersey
  - Merz Investigational Site #001207, Plainview, New York
  - Merz Investigational Site #001009, Winston-Salem, North Carolina
  - Merz Investigational Site #001206, Nashville, Tennessee
  - Merz Investigational Site #001183, Houston, Texas
- Canada (2):
  - Merz Investigational Site #001204, Halifax, Nova Scotia
  - Merz Investigational Site #001202, Winnipeg
- Czechia (4):
  - Merz Investigational Site #420024, Ostrava-Poruba
  - Merz Investigational Site #420031, Ostrava-Vitkovice
  - Merz Investigational Site #420030, Prague
  - Merz Investigational Site #420047, Rychnov nad Kněžnou
- France (2):
  - Merz Investigational Site #033018, Garches
  - Merz Investigational Site #033024, Rennes
- Germany (8):
  - Merz Investigational Site #049022, Beelitz-Heilstätten
  - Merz Investigational Site #049071, Düsseldorf
  - Merz Investigational Site #049079, Hamburg
  - Merz Investigational Site #049304, Kiel
  - Merz Investigational Site #049072, München
  - Merz Investigational Site #049148, München
  - Merz Investigational Site #049303, Regensburg
  - Merz Investigational Site #049302, Würzburg
- Italy (3):
  - Merz Investigational Site #039006, Messina
  - Merz Investigational Site #039011, Roma
  - Merz Investigational Site #039012, Roma
- Poland (13):
  - Merz Investigational Site #048057, Gdansk
  - Merz Investigational Site #048044, Kielce
  - Merz Investigational Site #048080, Krakow
  - Merz Investigational Site #048054, Krakow
  - Merz Investigational Site #048031, Krakow
  - Merz Investigational Site #048022, Lodz
  - Merz Investigational Site #048051, Lublin
  - Merz Investigational Site #048053, Poznan
  - Merz Investigational Site #048081, Poznan
  - Merz Investigational Site #048055, Warsaw
  - Merz Investigational Site #048023, Warsaw
  - Merz Investigational Site #048056, Warsaw
  - Merz Investigational Site #048033, Warsaw
- Russia (4):
  - Merz Investigational Site #007010, Krasnoyarsk
  - Merz Investigational Site #007011, Moscow
  - Merz Investigational Site #007009, Saint Petersburg
  - Merz Investigational Site #007012, Stavropol
- Spain (5):
  - Merz Investigational Site #034027, Madrid
  - Merz Investigational Site #034028, Majadahonda
  - Merz Investigational Site #034026, Seville
  - Merz Investigational Site #034030, Seville
  - Merz Investigational Site #034029, Terrassa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 331 individuals suffering from post-stroke lower-limb spasticity were screened and 290 were included in study at 51 sites. One ineligible subject was randomized to placebo but withdrawn from study prior to first treatment with study medication. For purpose of study analysis overall number of subjects enrolled is therefore considered 289.
Pre-assignment Details: A total of 290 subjects were enrolled in study. One ineligible subject was randomized to placebo but withdrawn from study prior to first treatment with study medication. A total of 289 subjects were enrolled in main period. All of the 269 subjects who completed the main period of the study entered the open-label extension period.
Groups:
- IncobotulinumtoxinA (Xeomin) 400 Units: IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  IncobotulinumtoxinA (400 Units): Main period: One injection session of solution, prepared by reconstitution of powder with 0.9 percent (%) Sodium Chloride (NaCl), 400 units, total volume 8.0 milliliter (mL); Mode of administration: intramuscular injection.
  IncobotulinumtoxinA (400 Units): Open-Label Extension Period: All subjects receive three injection sessions of solution, prepared by reconstitution of powder with 0.9% NaCl, 400 units, total volume 8.0 mL; Mode of administration: intramuscular injection.
- Placebo: Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection.
  Placebo Comparator: Main period: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding total placebo volume 8.0 mL; Mode of administration: intramuscular injection
Period: Main Period
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Started | 144 | 145
Treated | 144 | 145
Completed | 129 | 140
Not Completed | 15 | 5
Not completed — Death | 0 | 1
Not completed — Adverse Event | 6 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Predefined discontinuation criteria | 2 | 1
Period: Open-Label Extension Period
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Started | 269 | 0
Treated | 269 | 0
Completed | 218 | 0
Not Completed | 51 | 0
Not completed — Adverse Event | 15 | 0
Not completed — Withdrawal by Subject | 14 | 0
Not completed — Lack of Efficacy | 5 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance | 9 | 0
Not completed — Predefined discontinuation criteria | 6 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Evaluation Set (SES) is the subset of all subjects who were exposed to Investigational product (IP) in the main period at least once.
Groups:
- Main Period: IncobotulinumtoxinA (Xeomin) 400 Units: IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  IncobotulinumtoxinA (400 Units): Main period: One injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400 units, total volume 8.0 mL; Mode of administration: intramuscular injection.
- Main Period: Placebo: Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection.
  Placebo Comparator: Main period: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding total placebo volume 8.0 mL; Mode of administration: intramuscular injection
- Total: Total of all reporting groups
Arm/Group | Main Period: IncobotulinumtoxinA (Xeomin) 400 Units | Main Period: Placebo | Total
Number analyzed (Participants) | 144 | 145 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.2) | 57.0 (13.0) | 57.2 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 40 | 55 | 95
  Male | 104 | 90 | 194

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ashworth Scale (AS) for Plantar Flexors at Week 4
Description: The AS is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline and Week 4
Population: The Full Analysis Set (FAS) included subjects in the Safety Evaluation Set (SES) of the main period for whom the primary efficacy variable was available, whereby SES is the subset of all subjects who were exposed to IP in the main period at least once.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Number analyzed (Participants) | 144 | 145
Units on a scale
  Baseline | 2.8 (0.7) | 2.8 (0.7)
  Change at Week 4 | -0.4 (0.7) | -0.4 (0.7)
Statistical Analysis 1: Comparison: IncobotulinumtoxinA (Xeomin) 400 Units vs Placebo; The number of subjects included in the MMRM analysis was only 286 because a covariate was missing for 3 subjects; Test type: Superiority or Other; p = 0.777, Mixed-Model Repeated Measures; Least Square Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2]

2. Primary Outcome: Co-primary Variable: Investigator's Global Assessment of Efficacy at Week 12
Description: A 4-point Likert scale will be used with the ratings 1 = very good, 2 = good, 3 = moderate, and 4 = poor. Investigator's Global Assessment of Efficacy at Week 12 will be a co-primary outcome measure to fulfill post marketing commitments for U.S. regulatory authorities only. Elsewhere, it will be a secondary outcome measure.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Number analyzed (Participants) | 144 | 145
Percentage of Participants
  Very good | 3.5 | 4.8
  Good | 28.5 | 22.8
  Moderate | 22.2 | 26.9
  Poor | 45.8 | 45.5
Statistical Analysis 1: Comparison: IncobotulinumtoxinA (Xeomin) 400 Units vs Placebo; The statistical analysis provided was for all categories of this outcome measure; Test type: Superiority or Other; p = 0.804, Wilcoxon's Rank-Sum Test — worst-case analysis

3. Secondary Outcome: Response Rate for Plantar Flexors at All Post-Baseline Visits for Subjects With an Improvement (Reduction) of at Least 1 Point From Baseline in the Ashworth Scale (AS)
Description: Response is defined as an improvement (reduction) of the plantar flexor Ashworth Score by at least one score point. The AS is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Week 4, 8, and 12
Population: The FAS included subjects in SES of main period for whom primary efficacy variable was available, whereby SES is subset of all subjects who were exposed to IP in main period at least once. Here, "N"(Number of Participants Analyzed) and "n" signifies those participants who were evaluable for this outcome measure and at given time point respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Number analyzed (Participants) | 142 | 144
Percentage of Participants
  Week 4 (n=142, 144) | 37.3 | 35.4
  Week 8 (n=140, 142) | 39.3 | 33.8
  Week 12 (n=135, 141) | 20 | 17
Statistical Analysis 1: Comparison: IncobotulinumtoxinA (Xeomin) 400 Units vs Placebo; Week 4. Number of subjects included in analysis was three less than the observed cases because of a missing covariate for the logistic regression analysis, that is, n=283 for week 4; Test type: Superiority or Other; p = 0.845, Regression, Logistic — observed cases analysis; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.63 to 1.74]
Statistical Analysis 2: Comparison: IncobotulinumtoxinA (Xeomin) 400 Units vs Placebo; Week 8. Number of subjects included in analysis was three less than the observed cases because of a missing covariate for the logistic regression analysis, that is, n=279 for week 8; Test type: Superiority or Other; p = 0.437, Regression, Logistic — observed cases analysis; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.73 to 2.04]
Statistical Analysis 3: Comparison: IncobotulinumtoxinA (Xeomin) 400 Units vs Placebo; Week 12. Number of subjects included in analysis was three less than the observed cases because of a missing covariate for the logistic regression analysis, that is, n=273 for week 12; Test type: Superiority or Other; p = 0.698, Regression, Logistic — observed cases analysis; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.59 to 2.21]

4. Secondary Outcome: Ashworth Scale (AS) for Plantar Flexors at All Post-Baseline Visits
Description: The AS is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension). Here, 'n' specifies those subjects who were evaluated for this outcome measure at given time point.
Time Frame: Baseline, Week 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin) 400 Units | Placebo
Number analyzed (Participants) | 144 | 145
Units on a scale
  Baseline (n=144, 145) | 2.8 (0.7) | 2.8 (0.7)
  Week 4 (n= 142, 144) | 2.4 (0.9) | 2.4 (0.8)
  Week 8 (n=140, 142) | 2.4 (0.9) | 2.5 (0.7)
  Week 12 (n= 135, 141) | 2.7 (0.8) | 2.7 (0.7)

ADVERSE EVENTS:
Time Frame: From time point of first injection until 120 +/- 7 days after last administration of injection
Description: The investigator asked the subject for adverse events systematically at each visit.
Groups:
- Open-Label Extension: IncobotulinumtoxinA (Xeomin) 400 Units: IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  IncobotulinumtoxinA (400 Units): Open-Label Extension Period: All subjects receive three injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400 units, total volume 8.0 mL; Mode of administration: intramuscular injection.
Arm/Group | Main Period: IncobotulinumtoxinA (Xeomin) 400 Units | Main Period: Placebo | Open-Label Extension: IncobotulinumtoxinA (Xeomin) 400 Units
Serious Adverse Events (participants affected / at risk) | 6/144 | 5/145 | 22/269
Other Adverse Events (participants affected / at risk) | 13/144 | 13/145 | 31/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: IncobotulinumtoxinA (Xeomin) 400 Units (N=144) | Main Period: Placebo (N=145) | Open-Label Extension: IncobotulinumtoxinA (Xeomin) 400 Units (N=269)
Epilepsy (Nervous system disorders) | 1 | 0 | 2
Intracranial haematoma (Nervous system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cranioplasty (Surgical and medical procedures) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Medical induction of coma (Surgical and medical procedures) | 0 | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 0 | 0 | 1
Tracheostomy (Surgical and medical procedures) | 0 | 0 | 1
Limb operation (Surgical and medical procedures) | 0 | 0 | 1
Rehabilitation therapy (Surgical and medical procedures) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper-limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Immobile (Social circumstances) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Period: IncobotulinumtoxinA (Xeomin) 400 Units (N=144) | Main Period: Placebo (N=145) | Open-Label Extension: IncobotulinumtoxinA (Xeomin) 400 Units (N=269)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (9) | 10 (10)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (5)
Vision blurred (Eye disorders) | 3 (4) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 11 (12)
γ-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 7 (7)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the Investigator will consider these doubts in the publication as long as the scientific neutrality is not affected.